CLINICAL TRIAL: NCT00775216
Title: Project Diabetes: Prescription for Healthy Living
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: grant funding ended and lack of sufficient participants to complete trial
Sponsor: Vanderbilt University (Other)
Responsible Party: Bettina M. Beech, DrPH, MPH, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 080811
Record Dates: First submitted 2008-10-07; First posted 2008-10-20 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes Mellitus; Exercise; Obesity; Behavioral Research
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Obesity | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (No Intervention): Standard behavioral counseling
- Intervention (Experimental): Behavioral counseling intervention augmented with an interactive health promotion "telephone helpline"
  Interventions: Behavioral: Behavioral counseling plus "telephone helpline"

INTERVENTIONS:
Behavioral: Behavioral counseling plus "telephone helpline" — A trained behavioral counselor will place phone calls to Phase 2 intervention participants. These calls will be used to provide tailored physical activity advice and to extend our partnership with the Metro Nashville Parks and Recreation Department, directing participants to community centers close to their homes or workplaces where they can access a variety of physical activities (e.g., indoor pools, walking tracks, fitness centers, greenways, etc) using a newly developed electronic database. Following an orientation to the Metro Parks services which will be held at either Hadley Regional Park or Coleman Regional Park, participants will be directed to the Metro Parks facility most convenient to them.
  Arms: Intervention

SUMMARY:
Health disparities related to obesity, pre-diabetes and Type 2 diabetes in the United States represent public health concerns. Given the benefit of exercise in disease prevention and management, evidence-based, cost-effective, brief interventions are needed to improve patient outcomes related to Type 2 diabetes and associated conditions. This novel behavioral intervention study connects individuals with resources within their community to affect change in their health and wellness. The aim is to connect disparate individuals to health and wellness resources to prevent the onset of diabetes. This will be accomplished through a collaborative effort with Vanderbilt Diabetes Center, Nashville Metro Parks and Recreation, and the Metro Public Health Department.

A time series design will be used to assess the efficacy of physical activity counseling delivered by a health care professional, plus continued contact intervention delivered via a proactive and reactive health promotion counseling hotline that will leverage our partnership with Metro Parks versus counseling advice alone. In order to refine this intervention (Phase II) before it is executed, focus groups will first be conducted in Phase I with members of the target population in order to obtain feedback on the proposed intervention activities and materials. Qualitative findings and feasibility testing will be the basis for modifying the intervention.

DETAILED DESCRIPTION:
Lifestyle changes, such as moderate physical activity (e.g. brisk walking) have been shown to delay or prevent the development of Type 2 diabetes in patients with obesity and pre-diabetes. Given the clear benefit of exercise in disease prevention and management, evidence-based cost-effective brief interventions are needed to improve patient outcomes related to Type 2 diabetes and associated health disparities.

In America over the last two decades, adult obesity rates have doubled from 15% to 30%. In 1990, no state had an obesity rate over 14%. In 2003, thirty-five states posted obesity rates of over 20%. Tennessee currently ranks fifth in the U.S. for highest rate of adult obesity. In 2003, direct medical costs associated with obesity totaled an estimated $1.84 billion in Tennessee. Medicare ($433 million) and Medicaid ($488 million) absorbed approximately 50% of these medical costs. Obesity is closely linked with such diseases as heart disease, stroke, diabetes, and certain cancers. In both East and South Nashville, cancer, heart disease, and stroke are listed as three of the top five causes of death with significant racial, educational, and economic disparities.

Reducing socioeconomic and racial/ethnic disparities in Type 2 diabetes among adults will require multiple interventions society-wide in order to provide cumulative and synergistic effects that can result in sustained health practices and improved patient outcomes. One step in this approach is to encourage health care providers to deliver health promotion advice and counseling to their patients during routine office visits. Another is to link advice with readily available resources wherein an individual might be able to implement counsel. Therefore, the specific aim of this proposal is to evaluate the relative contribution of a multi-component, behavioral counseling intervention delivered by health care professionals versus the same behavioral counseling intervention when augmented by an interactive health promotion "telephone helpline" that will, among other things offer guidance on the availability of physical activity resources at Metro Parks facilities. In order to refine this intervention (Phase II) before it is executed, focus groups will first be conducted in Phase I with members of the target population in order to obtain feedback on the proposed intervention activities and materials. Qualitative findings and feasibility testing will be the basis for modifying the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years old
* Overweight (BMI greater than or equal to 25)
* Sedentary (self-report less than 30 minutes of moderate physical activity most days of the week)
* Has a family member (parent, grandparent, or sibling) with diabetes or pre-diabetes

Exclusion Criteria:

* Participants unable to engage in physical activity (oxygen dependent, wheel chair bound, amputations, Class 3 or 4 NY Heart Association classification for Congestive Heart Failure)
* Non-English speaking

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be assessed by the short version of the International Physical Activity Questionnaire and the 6-minute Walk Test. | Baseline and 6 months

SECONDARY OUTCOMES:
Questions regarding readiness to change, self-efficacy, knowledge of and access to physical activity centers, basic demographics, height/weight, and blood pressure will be assessed. | Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bettina M. Beech, DrPH, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States